CLINICAL TRIAL: NCT04588246
Title: Phase III Trial of Stereotactic Radiosurgery (SRS) or Hippocampal-Avoidant Whole Brain Radiotherapy (HA-WBRT) for Distant Brain Relapse With Brain Metastasis Velocity >/= 4 Brain Metastases/Year
Brief Title: Comparing Whole Brain Radiotherapy Using a Technique That Avoids the Hippocampus to Stereotactic Radiosurgery in Patients With Cancer That Has Spread to the Brain and Come Back in Other Areas of the Brain After Earlier Stereotactic Radiosurgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRG-BN009; NCI-2020-07375 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BN009; NRG-BN009 (Other: NRG Oncology); NRG-BN009 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-04

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Lung Small Cell Carcinoma; Metastatic Malignant Breast Neoplasm; Metastatic Malignant Digestive System Neoplasm; Metastatic Malignant Neoplasm in the Brain; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Metastatic Renal Cell Carcinoma; Recurrent Brain Neoplasm; Stage IV Lung Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Breast Neoplasms; Gastrointestinal Neoplasms; Brain Neoplasms; Neoplasm Metastasis; Melanoma; Carcinoma, Renal Cell; Lung Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Memantine; Radiosurgery

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (memantine, HA-WBRT) (Experimental): Patients undergo HA-WBRT daily (5 times weekly) for 2 weeks for a total of 10 fractions in the absence of disease progression or unacceptable toxicity. Prior to HA-WBRT or no later than the 4th treatment, patients also receive memantine PO QD or BID for 24 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI and may undergo blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Memantine; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Whole-Brain Radiotherapy
- Arm II (SRS/fSRS) (Active Comparator): Patients undergo single fraction SRS or fSRS on study. Patients also undergo CT and MRI and may undergo blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Memantine — Given PO
  Arms: Arm I (memantine, HA-WBRT)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Radiosurgery — Undergo SRS/fSRS
  Other Names: SRS; Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
  Arms: Arm II (SRS/fSRS)
Radiation: Whole-Brain Radiotherapy — Undergo HA-WBRT
  Other Names: WBRT; whole-brain radiation therapy
  Arms: Arm I (memantine, HA-WBRT)

SUMMARY:
This phase III trial compares the effect of adding whole brain radiotherapy with hippocampal avoidance and memantine versus stereotactic radiosurgery alone in treating patients with cancer that has spread to the brain and come back in other areas of the brain after earlier stereotactic radiosurgery. Hippocampus avoidance during whole-brain radiation therapy decreases the amount of radiation that is delivered to the hippocampus, which is a brain structure that is important for memory. The medicine memantine is also often given with whole brain radiation therapy because it may decrease the risk of side effects of radiation on neurocognitive function (including thinking and memory). Stereotactic radiosurgery delivers a high dose of radiation only to the small areas of cancer in the brain and avoids the surrounding normal brain tissue. Adding whole brain radiotherapy with hippocampal avoidance and memantine may be effective in reducing the size of the cancer or keeping the cancer the same size when it has spread to the brain and/or come back in other areas of the brain compared to stereotactic radiosurgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if hippocampal-avoidant plus whole brain radiotherapy (HA-WBRT) in patients with distant brain failure with brain metastasis velocity >= 4 new brain metastases/year prolongs time to neurologic death as compared to stereotactic radiosurgery (SRS).

SECONDARY OBJECTIVES:

I. To determine if HA-WBRT in patients with distant brain failure with brain metastasis velocity >= 4 new brain metastases/year prolongs overall survival as compared to SRS.

II. To evaluate if HA-WBRT in patients with distant brain failure with brain metastasis velocity >= 4 new brain metastases/year prolongs intracranial progression-free survival as compared to SRS.

III. To evaluate if HA-WBRT in patients with distant brain failure with brain metastasis velocity >= 4 new brain metastases/year improves brain metastasis velocity at subsequent relapse as compared to SRS.

IV. To assess perceived difficulties in cognitive abilities, symptom burden and health status after HA-WBRT, as compared to SRS, in patients with distant brain failure with brain metastasis velocity >= 4 new brain metastases/year.

V. To compare neurocognitive function outcomes following HA-WBRT, as compared to SRS, in patients with distant brain failure with brain metastasis velocity >= 4 new brain metastases/year.

VI. To tabulate and descriptively compare the adverse events associated with the interventions.

VII. To tabulate and descriptively compare the number of salvage procedures used to manage recurrent intracranial disease following the interventions.

EXPLORATORY OBJECTIVES:

I. To collect serum, plasma, and whole blood for translational research analyses.

II. To collect baseline and all follow-up magnetic resonance (MR) imaging for hippocampal volume, memory center substructures, axial T2 volumes, and quantitative texture analysis.

III. To collect baseline and follow-up MR imaging to extract whole brain volume, white matter volume and volume of metastatic disease to correlate with cognitive change at 4 months.

IV. To evaluate dose-volume histogram parameters to correlate with radiation toxicity.

V. To assess in patients receiving immunotherapy or targeted therapy, if HA-WBRT in patients with distant brain failure with brain metastasis velocity >= 4 new brain metastases/year at time improves brain metastasis velocity and/or overall survival at subsequent relapse as compared to SRS.

VI. To compare the estimated cost of brain-related therapies and quality-adjusted life years in patients who receive HA-WBRT, as compared to SRS, in patients with distant brain failure with metastasis velocity >= 4 new brain metastases/year.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo HA-WBRT daily (5 times weekly) for 2 weeks for a total of 10 fractions in the absence of disease progression or unacceptable toxicity. Prior to HA-WBRT or no later than the 4th treatment, patients also receive memantine orally (PO) once daily (QD) or twice daily (BID) for 24 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and magnetic resonance imaging (MRI) and may undergo blood sample collection throughout the trial.

ARM II: Patients undergo single fraction SRS or fractionated SRS (fSRS) on study. Patients also undergo CT and MRI and may undergo blood sample collection throughout the trial.

Patients are followed up at 2, 4, 6, 9, and 12 months from the start of SRS/fSFS or HA-WBRT and then every 6 months after month 12 and within 21 days after patient death.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have developed their distant brain relapse(s) at least 8 weeks after last SRS and within 21 days prior to randomization

  * Distant brain relapse lesions to be treated must measure =< 3.0 cm in maximal extent and total volume of distant brain relapses to be treated must measure < 30 mL on the contrast-enhanced diagnostic MRI brain scan obtained within 21 days prior to randomization
  * "last SRS" refers to the most recent SRS procedure that the patient received prior to enrollment on this study
  * Distant brain relapse lesions must be diagnosed on MRI, which will include the following elements:

    * REQUIRED MRI ELEMENTS

      * Post gadolinium contrast-enhanced T1-weighted three-dimensional (3D) spoiled gradient (SPGR). Acceptable 3D SPGR sequences include magnetization-prepared 3D gradient recalled echo (GRE) rapid gradient echo (MP-RAGE), turbo field echo (TFE) MRI, BRAVO (brain volume imaging) or 3D fast FE (field echo). The T1-weighted 3D scan should use the smallest possible axial slice thickness, not to exceed 1.5 mm
      * Pre-contrast T1 weighted imaging (3D imaging sequence strongly encouraged)
      * A minimum of one axial T2 fluid attenuated inversion recovery (FLAIR) (preferred) or T2 sequence is required. This can be acquired as a 2D or 3D image. If 2D, the images should be obtained in the axial plane
    * ADDITIONAL RECOMMENDATIONS

      * Recommendation is that an axial T2 FLAIR (preferred) sequence be performed instead of a T2 sequence
      * Recommendation is that that pre-contrast 3D T1 be performed with the same parameters as the post-contrast 3D T1
      * Recommendation is that imaging be performed on a 3 Tesla (3T) MRI
      * Recommendation is that the study participants be scanned on the same MRI instrument at each time point
      * Recommendation is that if additional sequences are obtained, these should meet the criteria outlined in Kaufmann et al., 2020
      * If additional sequences are obtained, total imaging time should not exceed 60 minutes
* Brain metastasis velocity (BMV) since last SRS must be >= 4 brain metastases/year
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry
* Pathologically (histologically or cytologically) proven diagnosis of small cell cancer, non-small cell lung cancer, melanoma, breast cancer, renal cell carcinoma, or gastrointestinal cancer within 10 years prior to randomization. If the original histologic proof of malignancy is greater than 10 years, then pathological (i.e., more recent) confirmation is required (e.g., from a systemic metastasis or brain metastasis)

  * Other histologies are not permitted
* History and physical examination within 28 days prior to randomization
* Age >= 18
* Karnofsky performance status of >= 70 within 28 days prior to randomization
* Calculated creatinine clearance (CrCl) >= 30 ml/min (within 28 days prior to randomization)
* Blood urea nitrogen (BUN) within 1.5 times the institutional upper limit of normal (ULN) (e.g., if the ULN is 20 mg/dL, then BUN up to 30 mg/dL is permitted) (within 28 days prior to randomization)
* Negative urine or serum pregnancy test (in women of childbearing potential) within 14 days prior to randomization

Exclusion Criteria:

* BMV >= 4 brain metastases/year at time of any SRS prior to enrollment.

  * Patients are permitted to have undergone multiple SRS treatments to different brain metastases so long as prior BMV has been less than 4 brain metastases/year
* Prior WBRT or prophylactic cranial irradiation
* Local relapse of metastasis previously treated with upfront SRS (i.e., relapse outside previously SRS-treated metastases is allowed)
* Brain metastases from primary germ cell tumor or lymphoma
* Definitive leptomeningeal metastasis
* Planned cytotoxic chemotherapy on the same day as SRS or HA-WBRT; concurrent immunotherapy is permitted
* Radiographic evidence of enlargement or other architectural distortion of the lateral ventricles, including placement of external ventricular drain or ventriculoperitoneal shunt
* Known history of demyelinating disease such as multiple sclerosis
* Inability to swallow pills
* Contraindication to MR imaging such as non-MR conditional implanted metal devices or unknown metallic foreign bodies, or contraindication to gadolinium contrast administration during MR imaging, such as anaphylactic allergy that cannot be adequately addressed with pre-contrast medications or acute kidney injury
* Contraindications to memantine, including:

  * Allergy, including prior allergic reaction to memantine
  * Intractable seizures on adequate anticonvulsive therapy-more than 1 seizure per month for the past 2 months
  * Current use of N-methyl-D-asparatate (NMDA) agonist
  * Current alcohol or drug abuse, which can exacerbate lethargy/dizziness with memantine
* Severe, active co-morbidity defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of randomization
  * Chronic obstructive pulmonary disease exacerbation or other acute respiratory illness precluding study therapy at the time of randomization
  * Severe hepatic disease defined as a diagnosis of Child-Pugh class B or C hepatic disease
  * Renal tubular acidosis or metabolic acidosis
  * Human immunodeficiency virus (HIV) positive with CD4 count < 200 cells/microliter. Note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count >= 200 cells/microliter within 30 days prior to randomization. Note also that HIV testing is not required for eligibility for this protocol
* Pregnant or lactating women, or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the medication and radiation involved in this study has unknown effects on the unborn fetus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinai Gondi, Principal Investigator — NRG Oncology
Locations (81):
- United States (79):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - City of Hope Corona, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope South Bay, Torrance, California
  - City of Hope Upland, Upland, California
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
- CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec, Canada
- Pamela Youde Nethersole Eastern Hospital, Chai Wan, Hong Kong

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Memantine, HA-WBRT): Patients undergo hippocampal-avoidant whole brain radiotherapy (HA-WBRT) daily (5 times weekly) for 2 weeks for a total 30 Gy in 10 fractions in the absence of disease progression or unacceptable toxicity. Consolidative stereotactic radiosurgery (SRS) boost following HA-WBRT is permitted during the follow-up period before progression. Prior to HA-WBRT or no later than the 4th treatment, patients also receive memantine target twice daily (BID) dose 20 mg/day or target extended-release dose 28 mg/day in the absence of disease progression or unacceptable toxicity.
- Arm II (SRS/fSRS): Patients undergo salvage SRS or fractionated stereotactic radiosurgery(fSRS).
Period: Overall Study
Arm/Group | Arm I (Memantine, HA-WBRT) | Arm II (SRS/fSRS)
Started (Randomized) | 10 | 9
Completed (Participants contributing data to results are considered to have completed the study.) | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Arm I (Memantine, HA-WBRT): Patients undergo HA-WBRT daily (5 times weekly) for 2 weeks for a total 30 Gy in 10 fractions in the absence of disease progression or unacceptable toxicity. Consolidative SRS boost following HA-WBRT is permitted during the follow-up period before progression. Prior to HA-WBRT or no later than the 4th treatment, patients also receive memantine target BID dose 20 mg/day or target extended-release dose 28mg/day in the absence of disease progression or unacceptable toxicity.
- Arm II (SRS/fSRS): Patients undergo salvage SRS or fSRS.
- Total: Total of all reporting groups
Arm/Group | Arm I (Memantine, HA-WBRT) | Arm II (SRS/fSRS) | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Median (Full Range); unit: years] | 63.5 [52 to 75] | 60 [56 to 75] | 63 [52 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 7 | 9 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Karnofsky performance status [Count of Participants; unit: Participants] — 70 = Cares for self, unable to carry on normal activity or to do active work; 80 = Normal activity with effort, some signs or symptoms of disease; 90 = Able to carry on normal activity, minor signs or symptoms of disease; 100 = Normal no complaints, no evidence of disease.
  Participants
    70 | 3 | 2 | 5
    80 | 3 | 4 | 7
    90 | 4 | 3 | 7
Brain Metastasis Velocity (BMV) [Count of Participants; unit: Participants] — BMV = [Total number of new brain metastases since last SRS]/[Time interval (in years) since upfront SRS]. "Last SRS" refers to the most recent SRS procedure that the participant received prior to enrollment on this study. It is calculated at the time of distant brain relapse after SRS. Higher BMV is associated with lower rates of survival and higher rates of neurologic death.
  Participants
    4 - 13 | 2 | 4 | 6
    >13 | 8 | 5 | 13
Is participant receiving immunotherapy? [Count of Participants; unit: Participants]
  No | 8 | 8 | 16
  Yes | 2 | 1 | 3
Diagnosis-specific graded prognostic assessment (DS-GPA) [Count of Participants; unit: Participants] — A tool used by healthcare professionals to estimate the survival of patients with brain metastases based on the prognostic factors of the primary cancer. It provides a score ranging from 0 (worst prognosis) to 4 (best prognosis).
  Participants
    0-2 | 9 | 6 | 15
    3-4 | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Neurologic Death
Description: Neurologic death defined as 1) Progressive neurologic decline or new neurologic symptoms/signs at time of death irrespective of status of extracranial disease OR 2) Death from inter-current disease in patients with severe neurologic dysfunction. Neurologic death rates were to be estimated using the cumulative incidence method, treating non-neurologic deaths as competing risks, and otherwise censoring participants alive at time of analysis. Analysis was to occur after 127 neurologic death events overall. The primary comparison of treatment arms would be a one-sided 0.05-level test for cause-specific hazard ratio (CHR) in a Cox proportional hazards model. Given the small number of participants due to early study closure, only the number of patients with neurologic death is reported and no statistical testing was done.
Time Frame: From baseline to neurologic death or last follow-up. Maximum follow-up at time of study termination was 29.7 months.
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Groups:
- Arm II (SRS/Fractionated Stereotactic Radiosurgery(fSRS)): Patients undergo salvage SRS or fSRS.
Arm/Group | Arm I (Memantine, HA-WBRT) | Arm II (SRS/Fractionated Stereotactic Radiosurgery(fSRS))
Number analyzed (Participants) | 10 | 9
Participants | 3 | 3

2. Secondary Outcome: Overall Survival
Description: Survival rates were to be estimated using the Kaplan-Meier method and the treatment arms were to be compared using a stratified log-rank test. Given the small number of participants due to early study closure, only the number of patients alive at time of study termination is reported, and no statistical testing was done.
Time Frame: Baseline to death or last follow-up. Maximum follow-up at time of study termination was 29.7 months.
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Memantine, HA-WBRT): Patients undergo HA-WBRT daily (5 times weekly) for 2 weeks for a total 30 Gy in 10 fractions in the absence of disease progression or unacceptable toxicity. Consolidative SRS boost following HA-WBRT is permitted during the follow-up period before progression. Prior to HA-WBRT or no later than the 4th treatment, patients also receive memantine target BID dose 20 mg/day or target extended-release dose 28 mg/day in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I (Memantine, HA-WBRT) | Arm II (SRS/fSRS)
Number analyzed (Participants) | 10 | 9
Participants | 5 | 5

3. Secondary Outcome: Intracranial Progression-Free Survival (IPFS)
Description: IPFS rates were to be estimated using the Kaplan-Meier method and the treatment arms were to be compared using a stratified log-rank test. Given the small number of participants due to early study closure, only the number of patients with alive without intracranial progression is reported, and no statistical testing was done. Per the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria, intracranial progression is defined as local progression of lesions treated with prior radiation or distant progression/development of a new brain lesion. Given the small number of participants due to early study closure, only the number of patients alive without intracranial progression is reported and no statistical testing was done.
Time Frame: Baseline to intracranial progression, death, or last follow-up. Maximum follow-up at time of study termination was 29.7 months.
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Memantine, HA-WBRT) | Arm II (SRS/fSRS)
Number analyzed (Participants) | 10 | 9
Participants | 5 | 2

4. Secondary Outcome: Brain Metastasis Velocity at Subsequent Relapse (BMVs)
Description: BMVs = [total number of new brain metastases since on-study SRS/HA-WBRT] / (years since on-study SRS/HA-WBRT). BMVs is calculated at the time of distant brain relapse. Higher BMVs is associated with lower rates of survival and higher rates of neurologic death.
Time Frame: Baseline to death or last follow-up. Maximum follow-up at time of study termination was 29.7 months.
Population: Randomized participants who subsequently relapsed with new brain metastases
Measure: Median (Full Range); unit: brain metastases/year
Arm/Group | Arm I (Memantine, HA-WBRT) | Arm II (SRS/fSRS)
Number analyzed (Participants) | 0 | 5
brain metastases/year |  | 33.18 [21.90 to 104.29]

5. Secondary Outcome: Change From Baseline in the M.D. Anderson Symptom Inventory Brain Tumor Module (MDASI-BT) Symptom Severity Score
Description: The MD Anderson Symptom Inventory for brain tumor (MDASI-BT) is a 28-item multi-symptom patient-reported outcome measure assessing the presence and severity of symptoms experienced by cancer patients and the interference with daily living caused by these symptoms, with 9 items specific to brain tumors. Each item ranges from 0 ("not present") to 10 ("as bad as you can imagine") and is rated as the worst occurrence in the last 24 hours. The Symptom Severity subscale score is the average of the symptom severity items, ranging from 0 (best) to 10 (worst). Change from baseline is calculated as score at 4 months minus score at baseline. A negative change value indicates improvement in symptom severity, while a positive change value indicates worsening.
Time Frame: Baseline and 4 months from treatment start
Population: Randomized participants with data at baseline and 4 months from start of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Memantine, HA-WBRT) | Arm II (SRS/fSRS)
Number analyzed (Participants) | 5 | 4
score on a scale | -0.82 (1.29) | 0.53 (1.61)

6. Secondary Outcome: Number of Participants With a Grade 3 or Higher Adverse Event
Description: Common Terminology Criteria for Adverse Events (version 5.0) grades adverse event severity as follows: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = death related to adverse event. Adverse events reported as possibly, probably, or definitely related to treatment are considered to be treatment-related adverse events. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: Baseline to last follow-up. Maximum follow-up at time of study termination was 29.7 months.
Population: Randomized participants who started treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Memantine, HA-WBRT) | Arm II (SRS/fSRS)
Number analyzed (Participants) | 8 | 8
Participants | 4 | 3

7. Secondary Outcome: Number of Participants Who Received Salvage Procedures
Description: Salvage procedures are defined as procedures for the purpose of managing recurrent intracranial disease following protocol treatment.
Time Frame: Baseline to last follow-up. Maximum follow-up at time of study termination was 29.7 months.
Population: Randomized participants who started treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Memantine, HA-WBRT) | Arm II (SRS/fSRS)
Number analyzed (Participants) | 8 | 8
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Baseline to last follow-up. Maximum follow-up was 29.7 months.
Description: All-cause mortality was assessed in eligible participants. Adverse events were assessed in eligible participants who started protocol treatment.
Arm/Group | Arm I (Memantine, HA-WBRT) | Arm II (SRS/Fractionated Stereotactic Radiosurgery(fSRS))
All-Cause Mortality (participants affected / at risk) | 5/10 | 4/9
Serious Adverse Events (participants affected / at risk) | 4/8 | 1/8
Other Adverse Events (participants affected / at risk) | 6/8 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Memantine, HA-WBRT) (N=8) | Arm II (SRS/Fractionated Stereotactic Radiosurgery(fSRS)) (N=8)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Memantine, HA-WBRT) (N=8) | Arm II (SRS/Fractionated Stereotactic Radiosurgery(fSRS)) (N=8)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1
Blurred vision (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Floaters (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 3
Fever (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Weight loss (Investigations) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 1
Memory impairment (Nervous system disorders) | 4 | 0
Muscle weakness left-sided (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary urgency (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study stopped accrual and data collection early due to unmet targeted accrual goals, with 19 participants enrolled out of 350 planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT04588246/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT04588246/ICF_001.pdf